CLINICAL TRIAL: NCT02389036
Title: A Crossover, Cluster Randomised Controlled Trial of Selective Decontamination of the Digestive Tract in Intensive Care Unit Patients (SuDDICU)
Brief Title: Selective Decontamination of the Digestive Tract in Intensive Care Unit Patients
Acronym: SuDDICU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: Imperial College London (Other); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: GI-CCT070115
Record Dates: First submitted 2015-03-02; First posted 2015-03-17 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Critical Illness; Sepsis; Septic Shock; Ventilator Associated Pneumonia
MeSH Terms: conditions — Critical Illness; Sepsis; Shock, Septic; Pneumonia, Ventilator-Associated | interventions — Colistin; Tobramycin; Nystatin; Ceftriaxone; Cefotaxime; Ciprofloxacin

STUDY DESIGN:
Intervention Model Description: Cluster, crossover, randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group- standard care (No Intervention): Standard care- In Australia there are no national guidelines so local policy is determined by each ICU. We are recommending (but not mandating) that control and SDD group management be in line with these national guidelines. We will recommend control and SDD group management is in line with current national standards of practice that may or may not include a VAP bundle. We will monitor record data regarding the nature and delivery of the control and SDD group co-interventions.
- SDD intervention group (Experimental): The intervention will entail:
  1. A six-hourly topical application of 0.5g paste, containing colistin 10mg, tobramycin 10mg and nystatin 125,000 IU, to the buccal mucosa and oropharynx
  2. A six-hourly administration of 10 mL of a suspension containing 100 mg colistin, 80 mg tobramycin and 2 x 10^6 IU nystatin, to the gastrointestinal tract via a gastric/post-pyloric tube
  3. A four-day course of an IV antibiotic. Patients not already receiving a therapeutic antibiotic will be prescribed cefotaxime 1g six-hourly or ceftriaxone 1g daily, with dose adjusted as appropriate for organ dysfunction. Ciprofloxacin (400mg 12-hourly) may be used as an alternative if there is a contraindication to cephalosporins (e.g. allergy). Patients already receiving an alternative IV antibiotic to treat infection will not receive this additional IV antibiotic, but will continue the prescribed antibiotic for the usual duration of therapy.
  Interventions: Drug: SDD Oral Paste; Drug: SDD Gastric Suspension; Drug: Intravenous Antibiotic

INTERVENTIONS:
Drug: SDD Oral Paste — A six-hourly topical application of 0.5g paste, containing colistin 10mg, tobramycin 10mg and nystatin 125,000 IU, to the buccal mucosa and oropharynx
  Other Names: Colistin, Tobramycin and Nystatin
  Arms: SDD intervention group
Drug: SDD Gastric Suspension — 2. A six-hourly administration of 10 mL of a suspension containing 100 mg colistin, 80 mg tobramycin and 2 x 10 ^6 IU nystatin, to the gastrointestinal tract via a gastric/post-pyloric tube
  Other Names: Colistin, Tobramycin and Nystatin
  Arms: SDD intervention group
Drug: Intravenous Antibiotic — A four-day course of an intravenous antibiotic in patients not already receiving a therapeutic antibiotic
  Other Names: Ceftriaxone, Cefotaxime or Ciprofloxacin
  Arms: SDD intervention group

SUMMARY:
Introduction- Hospital acquired infections (HAI) are a major cause of morbidity and mortality and increase health care costs. Critically ill patients are particularly susceptible to these infections and have an even higher mortality. One intervention that has gained much interest in the medical literature for reducing infection rates and deaths from HAIs is selective decontamination of the digestive tract (SDD). SDD involves the application of antibiotic paste to the mouth, throat, stomach and a short course of intravenous antibiotics. The evidence supporting the use of SDD for saving lives and preventing infections is actually quite strong. However, health care professionals in many parts of the world have refrained from using SDD due to fears of the effects of overuse of antibiotics on the frequency of infections with resistant bacteria such as multi-resistant Gram negative organisms, MRSA and Clostridium difficile.

SuDDICU is a cross-over, cluster randomised trial comparing the effect of using selective decontamination of the digestive tract (SDD) plus standard care, to standard care alone on hospital mortality in patients receiving mechanical ventilation in the intensive care unit (ICU).

Secondary outcomes include an ecological assessment and a long-term health economic analysis.

DETAILED DESCRIPTION:
Design- international, multicentre, crossover, cluster randomised controlled trial (x-cRCT) of eligible patients in participating ICUs using two 12-month interventional trial periods separated by a 3-month inter-period gap.

An observational ecological assessment will be conducted in all ICU patients during one week of each month during the 3-month surveillance period before the first intervention period; in all trial eligible patients during the two 12-month intervention periods; in all ICU patients during one week of each month of the final 3-months of the two intervention periods; in all ICU patients during one week of each month during the 3-month inter-period and post-trial periods.

Participants- General ICUs that admit mechanically ventilated patients will be randomised in the first 12-month period to either implement the SDD protocol in addition to standard care or to continue standard care without SDD, and then to cross over to the other arm during the second 12-month period.

Eligible patients are defined as:

1. All patients who are mechanically ventilated via an endotracheal tube on admission to the ICU and who are predicted to remain ventilated beyond the end of the calendar day after the day of ICU admission, or
2. All patients who become mechanically ventilated via an endotracheal tube during their ICU stay and who are predicted to remain ventilated beyond the end of the calendar day after the day they are first ventilated, or
3. All patients who not already recruited but are receiving mechanical ventilation via an endotracheal tube and are expected to receive ongoing ventilation for a further 48-hours or more despite an earlier prediction that ventilation would be discontinued earlier.

All patients eligible for the intervention will receive the following in addition to the usual infection control measures:

1. 1. A six-hourly topical application of 0.5g paste, containing colistin 10mg, tobramycin 10mg and nystatin 125,000 IU, to the buccal mucosa and oropharynx
2. A six-hourly administration of 10 mL of a suspension containing 100 mg colistin, 80 mg tobramycin and 2 x 106 IU nystatin, to the gastrointestinal tract via a gastric/post-pyloric tube
3. A four-day course of an IV antibiotic. Patients not already receiving a therapeutic antibiotic will be prescribed cefotaxime 1g six-hourly or ceftriaxone 1g daily, with dose adjusted as appropriate for organ dysfunction. Ciprofloxacin (400mg 12-hourly) may be used as an alternative if there is a contraindication to cephalosporins (e.g. allergy). Patients already receiving an alternative IV antibiotic to treat infection will not receive this additional IV antibiotic, but will continue the prescribed antibiotic for the usual duration of therapy.

Statistical considerations and sample size- SuDDICU will recruit 10 000 to 15 000 patients from 29 ICUs and will have 80% power to detect an absolute reduction in hospital mortality of 3-5% from a baseline mortality of 29%, depending on the precise number of clusters.

ELIGIBILITY:
Inclusion Criteria:

Site inclusion for cluster study- A general ICU or complex of ICUs (medical, surgical, mixed) capable of treating mechanically ventilated critically ill adult patients.

Patient inclusion criteria

1. All patients who are mechanically ventilated via an endotracheal tube on admission to ICU and who are predicted to remain ventilated beyond the end of the calendar day after the day of ICU admission, or
2. All patients who become mechanically ventilated via an endotracheal tube during their ICU stay and who are predicted to remain ventilated beyond the end of the calendar day after the day they are first ventilated, or
3. All patients not already recruited who are receiving mechanical ventilation via an endotracheal tube and are expected to receive ongoing ventilation for a further 48 hours or more despite an earlier prediction that ventilation would be discontinued earlier.

Site exclusion criteria for cluster study-

1. Unwilling or unable to follow trial protocols.
2. Unable to capture the minimum data set required for the study.
3. Isolated specialty ICUs not co-located with a general ICU, such as solely cardiac, neurological/neurosurgical and burns ICUs, but such specialty patients cared for in general ICUs will be included
4. Specialty paediatric ICUs

Exclusion Criteria:

Patient exclusion criteria

1. Patients enrolled in a trial that would interact with the intervention
2. Patients with a known allergy, sensitivity or interaction to trial topical intervention drugs
3. Patients who are known or suspected to be pregnant
4. Patients who are moribund and not expected to survive the next 12 hours
5. Patients less than 16 years of age will not be enrolled in the UK

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20010 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Hospital Mortality | Hospital discharge [up to Day 90 after randomization]
  all-cause mortality at time of hospital discharge

SECONDARY OUTCOMES:
Total antibiotic usage | during ICU admission
  Total antibiotic usage (as daily defined doses) during ICU admission in all ICU admissions.
The incidence of antibiotic resistant organisms in cultures from blood or other sterile sites | during ICU admission
  The incidence of antibiotic resistant organisms in cultures from blood or other sterile sites during ICU admission in all ICU admissions.
The incidence of antibiotic-resistant organism in non-sterile clinical and surveillance specimens | during ICU admission
  The incidence of antibiotic-resistant organism in non-sterile clinical and surveillance specimens during ICU admission in all ICU admissions
The incidence of C. difficile infections | during ICU admission
  The incidence of C. difficile infections during ICU admission in all ICU admissions
Changes in antibiotic resistance rates between study epochs (pre-trial, interperiod gap and post-trial) within groups | Through out all study periods
  Changes in ARO rates between time epochs (pre-trial, trial, inter-period gap and post-trial) within groups. With control group data to give the secular trend in ARO with time and SDD group data studying the effects of SDD withdrawal from practice in the year after SDD delivery
Duration of mechanical ventilation | Time of enrolment to ICU discharge within index hospital admission,[up to Day 90 after randomization]
  Duration that the patient is mechanically ventilated in the ICU
ICU length of stay | From the time of enrolment to ICU discharge, [up to Day 90 after randomization]
  The length of time a patient stays in the ICU
Hospital length of stay | From time of enrolment to hospital discharge within the index hospital admission, [up to Day 90 after randomization]
  The total hospital length of stay for patient
ICU Mortality | ICU discharge [up to Day 90 after randomization]
  mortality at time of ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: John Myburgh, MBBCh PhD, Study Chair — The George Institute; Brian Cuthbertson, MD FRCA, Study Chair — Sunnybrook Health Sciences Centre; Anthony Gordon, MD FRCA, Study Chair — Imperial College London
Locations (3):
- The George Institute for Global Health, Sydney, New South Wales, Australia
- Sunnybrook Health Sciences Centre, Toronto, Canada
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The protocol and statistical analysis plan were made public in 2020. The participant level dataset will not be publicly available immediately but will be available to collaborative researchers after consultation and negotiation with the SuDDICU Investigators.
Supporting Information: Study Protocol, SAP
Time Frame: The SuDDICU Protocol V4.0 and SAP V1.1 are available on the open science framework in pre print.
Access Criteria: Public access, no access criteria to view the SuDDICU Protocol V4.0 and SAP V1.1
URL: https://osf.io/

REFERENCES:
- [Result] Cuthbertson BH, Campbell MK, MacLennan G, Duncan EM, Marshall AP, Wells EC, Prior ME, Todd L, Rose L, Seppelt IM, Bellingan G, Francis JJ. Clinical stakeholders' opinions on the use of selective decontamination of the digestive tract in critically ill patients in intensive care units: an international Delphi study. Crit Care. 2013 Nov 8;17(6):R266. doi: 10.1186/cc13096. PMID 24207137
- [Result] Daneman N, Sarwar S, Fowler RA, Cuthbertson BH; SuDDICU Canadian Study Group. Effect of selective decontamination on antimicrobial resistance in intensive care units: a systematic review and meta-analysis. Lancet Infect Dis. 2013 Apr;13(4):328-41. doi: 10.1016/S1473-3099(12)70322-5. Epub 2013 Jan 25. PMID 23352693
- [Result] Cuthbertson BH, Francis J, Campbell MK, MacIntyre L, Seppelt I, Grimshaw J; SuDDICU study groups. A study of the perceived risks, benefits and barriers to the use of SDD in adult critical care units (the SuDDICU study). Trials. 2010 Dec 3;11:117. doi: 10.1186/1745-6215-11-117. PMID 21129208
- [Derived] SuDDICU Investigators for the Australia and New Zealand Intensive Care Society Clinical Trials Group and the Canadian Critical Care Trials Group; Cuthbertson BH, Billot L, Campbell MK, Daneman N, Davis JS, Delaney A, Devaux A, Ferguson ND, Finfer SR, Fowler R, Gordon AC, Hammond NE, Klein G, Li Q, Marshall J, Micallef S, Murthy S, Mysore J, Naik C, Patel C, Pinto R, Rose L, Seppelt IM, Venkatesh B, Young PJ, Myburgh JA. Selective Decontamination of the Digestive Tract during Ventilation in the ICU. N Engl J Med. 2025 Oct 29. doi: 10.1056/NEJMoa2506398. Online ahead of print. PMID 41159880
- [Derived] Billot L, Cuthbertson B, Gordon A, Al-Beidh F, Correa M, Davis J, Finfer S, Glass P, Goodman F, Hammond N, Iredell J, Miller J, Murthy S, Rose L, Seppelt I, Taylor C, Young P, Myburgh J; SuDDICU Investigators. Protocol summary and statistical analysis plan for the Selective Decontamination of the Digestive Tract in Intensive Care Unit Patients (SuDDICU) crossover, cluster randomised controlled trial. Crit Care Resusc. 2023 Oct 18;23(2):183-193. doi: 10.51893/2021.2.oa5. eCollection 2021 Jun. PMID 38045525
- [Derived] Young PJ, Devaux A, Li Q, Billot L, Davis JS, Delaney A, Finfer SR, Hammond NE, Micallef S, Seppelt IM, Venkatesh B, Myburgh JA; SuDDICU Australia Investigators and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Selective digestive tract decontamination in critically ill adults with acute brain injuries: a post hoc analysis of a randomized clinical trial. Intensive Care Med. 2024 Jan;50(1):56-67. doi: 10.1007/s00134-023-07261-y. Epub 2023 Nov 20. PMID 37982826
- [Derived] SuDDICU Investigators for the Australian and New Zealand Intensive Care Society Clinical Trials Group; Myburgh JA, Seppelt IM, Goodman F, Billot L, Correa M, Davis JS, Gordon AC, Hammond NE, Iredell J, Li Q, Micallef S, Miller J, Mysore J, Taylor C, Young PJ, Cuthbertson BH, Finfer SR. Effect of Selective Decontamination of the Digestive Tract on Hospital Mortality in Critically Ill Patients Receiving Mechanical Ventilation: A Randomized Clinical Trial. JAMA. 2022 Nov 15;328(19):1911-1921. doi: 10.1001/jama.2022.17927. PMID 36286097